CLINICAL TRIAL: NCT01723033
Title: Differences in Cognitive Performance and Brain Activity Between Patients With PTSD and OCD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Doron Todder, Dr., Beersheva Mental Health Center
Other Study IDs: BHMC-5200
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: PTSD; OCD
Keywords: PTSD; OCD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- EEG acquisition: 15 PTSD patients and 15 OCD patients who will, while wearing a net of electrodes for EEG acquisition on their heads, perform three error detection tasks.
- Control: Previously collected healthy student's data

SUMMARY:
Comparison of the neurophysiological response of OCD and PTSD patients (both considered anxiety syndromes) in error processing. The patients will perform three computerized tasks while a net of electrodes (for EEG measurement) will be placed on their head. This data will then be compared to a previously collected healthy control sample.

DETAILED DESCRIPTION:
Scientific background Obsessive Compulsive Disorder (OCD) Obsessive Compulsive Disorder (OCD) is a chronic mental disturbance classified as an anxiety disorder, which causes a severe social and occupational damage. It is characterized with repetitive and intrusive thoughts, and with the urge to perform reoccurring rituals. Illness' course is usually chronic and is characterized with fluctuation in symptoms severity. Only a minority of patients gain full relief, even following the appropriate treatment. There are two main useful treatments, a behavioral therapy and a medicinal treatment using SSRI's. Even though medicinal treatments are improving, large amount of patients are irresponsive to a variety of medicinal treatment and about a third is classified as Refractory to Treatment. Of those who will gain relief, relapse rate is high (Catapano et al., 2006).

Brain imaging studies demonstrate that the neurophysiological basis of OCD appears to be abnormal functioning of frontal subcortical circuits and that illness' symptoms are related to an increase in cortical activity of different areas: anterior cingulate gyrus (Saxena & Rauch, 2000) orbitofrontal cortex, caudate nucleus, and thalamus. ERP studies provide a number of indicators of cerebral abnormalities in OCD, during critical aspects of cognitive processing (Clark et al., 2009). The sharp negative deflection associated with errors is referred to as error-related negativity (ERN; Gehring, Coles, Meyer, & Donchin, 1995). Gehring et al. (2000) found that OCD patients had an increased ERN amplitude which was significantly associated with symptom severity. Johannes et al. (2001) using a visual discrimination task also reported larger ERN amplitudes in OCD patients, whilst Hajcak and Simons (2002) found increased ERN-like deflections to both incorrect and correct trials in University under- graduates with high levels of obsessive compulsive characteristics.

From cognitive behavioral perspective, obsessive-compulsive disorder (OCD) has been associated with impairments in stop-signal inhibition, a measure of motor response suppression (Morein-Zamir, Fineberg, Robbins, & Sahakian, 2010). Another study has related OCD to an attention bias shifting towards the right hemifield in a well-established visual attention task (Maril, Hermesh, Gross-Isseroff, & Tomer, 2007). Furthermore this shift of attention had been reported to be positively correlated with OCD symptoms as measured by the Y-BOCS (e.g. less Y-BOCS score correlated with less shifting of attention).

Post-Traumatic Stress Disorder (PTSD) Posttraumatic stress disorder (PTSD) is associated with increased rates of health complaints (Beckham et al., 1998) medical morbidity (Beckham et al., 2003) health service utilization (Calhoun, et al., 2002), and mortality (Boscarino, 2006). The prevalence of PTSD in the general population is estimated to be between 7% and 12% (Breslau, 2009).

On the anatomical level reports vary with certain areas emerging as possibly implicated in PTSD predisposition and pathology. The hippocampus, important in learning and memory, has been shown to be reduced in volume in PTSD patients ( reviewed by Nutt & Malizia, 2004). Two additional regions implicated in PTSD are the amygdale- involved in emotional behavior, and the medial frontal cortex - important in regulation of the HPA axis ( reviewed by Nutt & Malizia, 2004).The major shortcoming of these anatomical studies is their retrospective nature, precluding the possibility of extracting causality. Thus the question of temporal sequence remains to be resolved.

Data reviewed by Etkin et al. (2011) suggest a controlled conscious top-down regulation, like emotional conflict regulation, uses ventral ACC and mPFC areas to inhibit negative emotional processing in the amygdala, thus dampening task interference. The ventral ACC and mPFC might thus perform a generic negative emotion inhibitory function that can be recruited by other regions (e.g. dorsal ACC and mPFC and lateral PFC) when there is a need to suppress limbic reactivity. One might speculate that a dysfunction in this circuit might contribute to a PTSD dysfunction in regulating negative emotional conflict. Unable to regulate and suppress emotional arousal related to trauma relevant information, the PTSD affected individual might choose to avoid it all together. The limbic reactivity might contribute to hyper vigilant responses, and affect memory processes leading to intrusion, as well. In short, dysfunction in the ventral medial PFC structures and their connections might contribute to all symptom clusters.

Summary Taken together the described neurophysiological and neuropsychological findings, it is compelling to further investigate antinational and response inhibition mechanisms in OCD patients compared to PTSD patients by tapping on performance in cognitive paradigms sensitive to the activity in medial prefrontal brain structures.

Study goal This study's main goal is to compare OCD and PTSD which are both considered an anxiety syndrome by means of the patient's performance and neurophysiologic response while engaged in an error detection task.

Design For the primary goal of the study, we will use a cross section design by comparing PTSD sample to the OCD sample. Cognitive and electrophysiological data from the clinical population will be compared to a previously collected healthy student's data.

Protocol After an explanation of the required procedure, all subjects will be kindly asked to sign an informed consent version that can be found on the ethics committee application form. Depicted in Figure 1, psychiatric and neurocognitive assessments will be taken at the clinical neurophysiology department at the Beer-Sheva Mental Health Institute and cognitive tasks while recording electrophysiology data will take place at the Cognitive Neurophysiology Lab at Ben Gurion University of the Negev.

Figure 1

In order to evaluate the error processing in a domain general perspective, the electrophysiological research will include three computerized tasks. In all three procedures the subjects will be asked to perform a task, while a net of electrodes for EEG acquisition will be placed on their head. During all tasks a number of within task breaks are inserted in order to reduce the discomfort of the subjects as much as possible. The total procedure, including all tasks, breaks within and in between tasks, will require approximately 2 hours.

Task description:

1. The Attention network test (Fan, McCandliss, Sommer, Raz, & Posner, 2002) has been previously implemented in studying of clinical disorders (Posner & Rothbart, 2007). In this task subject will be presented with five horizontal arrow stimuli and will be asked to identify the direction of the centrally presented arrow by pressing a button with the index finger. The procedure will require approximately 30 minutes.
2. In the Stroop with misspelled words task (Mesika & Berger, in preparation) subjects will be asked to name the color of the word presented, while avoiding its meaning. On some trials, spelling errors will be inserted in the presented words, while in others no spelling errors will be present. This procedure will require approximately 30 minutes.
3. The Arithmetic verification task is a modified version of the task which Tzur and colleagues have used previously (Tzur, Berger, Luria, & Posner, 2010; Tzur & Berger, 2007). The subjects participating in the task will be presented with either correct (e.g. 3X6=18) or incorrect (e.g. 3X6=21) arithmetical equations, and will be asked to decide each trial whether the equation presented is correct or incorrect. This procedure will require approximately 45 minutes.

Three weeks after the initial examination, all subjects will be invited to participate in a follow-up session at the Cognitive Neurophysiology Lab at Ben Gurion University of the Negev regardless of the treatment they were participating in during this period. At this point all subjects will be kindly asked to sign a new informed consent so that there will be no obligatory relationship been participating at the first phase and at follow-up of the experiment. Also, the subject's treatment between the sessions will be determined by the patients attending physician without the intervention of the research team.

Patients will be evaluated using several widely used rating scales adminstered by a trained psychiatrist.

Neurocognitive assessment

1. Raven's Progressive Matrices (Raven, 2000) - a measure of fluid intelligence; a factor which may be relevant to PTSD development. This will also allow better control for differences between patients normal population.
2. MindStreams®: neurocognitive assessment battery. Regularly used for diagnostic purposes in the center.

All cognitive assignments are computerized and will take place at the Clinical Neurophysiology department at the Beer-Sheva Mental Health center. The patient will either read the instructions on the computer monitor or a trained experimenter will read the task instruction for him.

Electrophysiology data acquisition

EEG recordings will take place at both the initiation and at the end of the research protocol. We will use the EGI Geodesic Sensor net (128 electrodes) and system for data acquisition (Electrical Geodesics, Oregon, USA). All equipment and materials that will be used are FDA approved for clinical and research use and are been routinely applied on patients, children and infants therefore can be considered safe. During all procedures the use of the equipment will be according to the manufacturer's instructions only.

Before applying the net, subject's head will be measured in order to determine the appropriate net size for EEG recording. Afterwards, using a soft and wide edged china marker, a small mark will be drawn on the scalp to indicate the midpoint of the head. While measuring the head, the electrode net will be dipped in electrolyte solution, composed of purified water, salt and baby shampoo. The solution then will be warmed up to body temperature to minimize the discomfort which could be caused by wetting the subject's head. During net application procedure no scraping of the scalp is required. Preparation process should take no more than 20 minutes and will cause no distress to the subject.

Statistics

Behavioral data will be collected as reaction time (in milliseconds) and accuracy (in proportion) for each condition for each task, and will be analyzed using analysis of variance (ANOVA) method for between subject analyses. Within subject analyses will be performed using the repeated measures ANOVA on the same variables.

EEG data will be analyzed using the event related potentials (ERP) method, extracting the amplitude (in microvolt) and latency (in milliseconds) of electrophysiological components. In the statistical analysis ANOVA and repeated measures ANOVA will be implemented accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD or OCD by DSM-IV criteria;
* For OCD subjects a Y-BOCS score larger than 16 composted form both obsession and compulsion patient's responses;
* For PTSD population a CAPS score larger than 40.
* Either no medicated patients or a combination of anti-anxiety, anti-depressant and tranquilizers.
* Patients with minimum depression symptoms (MDRAS < 18)

Exclusion Criteria:

* A medical history of other major psychiatric disorder.
* A known ailment of the central nervous system.
* No history of loss of consciousness.
* No history of head injury or abnormal head trauma upon routine imaging.
* No anti-psychotic or anti-epileptic and tricyclic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the outpatient clinic of the Beersheva Mental Health Center. 15 OCT and 15 PTSD patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (Y-BOCS)

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRAS)

OTHER OUTCOMES:
Clinician rating scale for assessing current and lifetime PTSD (CAPS)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Todder, MD, Principal Investigator — Beersheva Mental Health Center and Ben Gurion University of the Negev